CLINICAL TRIAL: NCT06379945
Title: Unified platforM for a Better integRal Evaluation of MyeLodyspLastic Syndromes in SpAin-Strategy for Unraveling Personalized genoMic Medicine in Public heAlth System (UMBRELLA-SUMMA)
Acronym: UMBRELLA-SUMMA
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI23/01103; PI2024 01 1484 (Registry Identifier: Ethics Committee for Drug Research of the Salamanca Health Area)
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Optical Genome Mapping; Next Generation Sequencing; Artificial Intelligence; Clonal evolution
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mononuclear cells, DNA, RNA and plasma from bone marrow and/or peripheral blood of MDS patients (MNC;MSC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myelodysplastic Syndromes (MDS) are heterogeneous clonal diseases characterized by difficult diagnosis, complex prognostic stratification and unsatisfactory treatment. Based on that, UMBRELLA SUMMA aims to provide better clinical management and personalized medicine to MDS patients in Spain through improving diagnosis (1), prognosis (2 and 3), and treatment (2), and facilitating future investigations (4) of the disease.

More concretely, we propose: 1. The application of new technologies such as Optical Genome Mapping (OGM) in the diagnosis of those MDS cases whose cytogenetic alterations cannot be identify by other methods, as well as the implementation of this technology using peripheral blood avoiding more invasive methods for patients. 2. To provide all Spanish Group of MDS (GESMD) members who require it with the newly prognostic stratification of their patients (IPSS-M) by making Next Generation Sequencing (NGS) accessible for all of them. 3. Validate and improve a new prognostic system (AIPSS-MDS) previously developed within the GESMD, thanks to artificial intelligence, one of the tools with the most projection in the field of medicine currently. 4. To build and register ISCIII collections of cells, genetic material and/or plasma from all prospective MDS patients.

On the other hand, the dynamics of coexisting mutations in a specific context of chromosomal abnormalities could be defining the clinical fate of each patient. Based on that, the IBSAL team recently proposed three models of MDS evolution based on NGS data from three different cytogenetic subgroups: normal karyotype, trisomy 8 and 5q deletion. The IBSAL proposal aims to deepen into the pathophysiological mechanisms of MDS evolution in these three models through in vitro and in vivo functional studies and single-cell multiomics approaches.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are hematologic malignancies characterized by bone marrow dysplasia, cytopenias (anemia, infections, bleeding), and a high risk of progression to acute myeloid leukemia (AML). Diagnosis and prognostic stratification are challenging, and treatment outcomes remain suboptimal, especially in elderly patients, who represent the majority of cases.

Beyond structural cytogenetic abnormalities found in 40-70% of patients, over 90% of MDS cases harbor somatic mutations impacting cellular function. Next-generation sequencing (NGS) has improved diagnosis, prognostication, and therapeutic decision-making.

The Spanish Group of MDS (GESMD) brings together over 400 professionals across 100+ centers and maintains RESMD, the world's largest MDS patient registry. In 2020, GESMD launched UMBRELLA to provide NGS access to participating centers, addressing a key clinical gap.

Building on UMBRELLA's success, the UMBRELLA-SUMMA project will:

1. Implement Optical Genome Mapping (OGM) to enhance detection of chromosomal alterations, especially in cases where standard cytogenetics fail. We will explore the use of peripheral blood samples to minimize invasiveness.
2. Expand access to NGS to GESMD members lacking this technology, supporting prognostic classification based on the IPSS-M, an updated molecularly integrated scoring system.
3. Apply Artificial Intelligence (AI) to validate and improve a new AI-driven prognostic model for MDS developed within GESMD.

Additionally, the project will create biobanks of biological samples from GESMD patients, linked to clinical and epidemiological data within RESMD, ensuring optimal and regulated access for future research.

Given MDS heterogeneity, personalized medicine is essential. UMBRELLA-SUMMA will address this through the study of different patient subgroups (low-risk, high-risk, AML-transformed MDS) with a multidisciplinary team comprising clinicians, biologists, biotechnologists, and bioinformaticians.

Results will be disseminated among healthcare professionals, patients and their families via GESMD's patient resources, institutional websites, social media, and public engagement activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients with a confirmed diagnosis of MDS by cytogenetics and/or morphological analysis
* Patients with complete clinical data
* Patients who sign the informed consent

Exclusion Criteria:

* Patients under 18 years old
* Patients who do not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myelodysplastic Syndrome at diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Structural variants and complex rearrangements in MDS | Baseline
  Optical Genome Mapping will be used to determine the presence of structural variant and complex rearrangements not detected by other conventional techniques
Mutations in MDS | Baseline and follow up
  Next Generation Sequencing will be use to define the IPSS-M (the International Molecular Prognostic Scoring System) in patients with MDS
Overall survival and leukemia-free survival in patients with MDS | Baseline
  The AIPSS-MDS (Artificial Intelligence Prognostic Scoring System for MDS) model will be validated to provide a personalized risk estimate for each individual patient
ISCIII collections of viable samples | Baseline
  To build and register ISCIII collections of viable samples (PB and BM cells), genetic material and/or plasma from all prospective MDS patients

CONTACTS AND LOCATIONS:
Overall Officials: María Díez Campelo, PhD MD, Study Chair — Instituto de Investigación Biomédica de Salamanca
Locations (4):
- Spain (4):
  - Fundación Instituto de Investigación Germans Trias i Puyol, Badalona, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Clínica Universitaria de Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided